CLINICAL TRIAL: NCT01367405
Title: COSMIC: Conservative or Early Surgical Management of Incomplete Cervical Cord Syndrome Without Spinal Instability. Randomized Controlled Trial
Brief Title: Comparing Surgical Decompression Versus Conservative Treatment in Incomplete Spinal Cord Injury
Acronym: COSMIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: only 1 inclusion in 1.5 years due to strict exclusion criteria
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL36977.091.11
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2013-11

CONDITIONS: Central Spinal Cord Syndrome
Keywords: Surgical decompression; conservative treatment; incomplete spinal cord lesion; recovery
MeSH Terms: conditions — Central Cord Syndrome | interventions — Decompression, Surgical; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgical decompression (Experimental): surgical decompression within 24 hours post-injury
  Interventions: Procedure: Surgical decompression
- Conservative treatment (Active Comparator): Normal conservative treatment without surgical intervention
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Surgical decompression — Surgical decompression within 24 hour postinjury
  Arms: surgical decompression
Procedure: Conservative treatment — Usual conservative treatment without surgery
  Arms: Conservative treatment

SUMMARY:
Traumatic Central Cord Syndrome (TCCS) was until recent recognized as a separate clinical entity. The most characteristic feature is the disproportionate more motor impairment of the arms and especially the hands than the legs, bladder dysfunction and sensory.

Recently, it has been shown that the distinction of TCCS with an incomplete cervical spinal cord lesion (ICSCL) is artificial. It is the most frequent incomplete traumatic spinal cord lesion. It accounts for up to 70 % of all incomplete cervical spinal cord lesions. The exact incidence is not known.

Uncertainty about the treatment exists. A good recovery has been described after conservative treatment. Conservative treatment was usually considered when a fracture or dislocation of the spine were absent. It is often seen in hyperextension trauma in the elderly with degenerative spondylotic stenotic cervical spine. However, some reports suggest a better outcome after surgical decompression. Randomized trials have not been performed. To avoid discussion about possible confounding or effect modification related to the mechanism of trauma, this study will focus on ICSCL in patients without fracture or instability of the cervical spine on radiological examination. Also the problem of crossover from the conservative group to the surgical one due to the nature of spinal instability will be reduced.

Goal of the study: To compare the efficacy of early decompressive surgery to improve functional outcome in patients with ICSCL without a fracture or instability of the cervical spine compared to those receiving conservative treatment.

Definition of ICSCL in this study: ICSCL is an incomplete spinal cord lesion due to a cervical spine trauma. At CT scanning with reconstruction and at MRI signs are not seen that could indicate a fracture of the cervical spine or instability. An overt sequestrated herniated disc should not be present since this will always necessitate immediate surgery. Involvement of the cervical spinal cord should be established at physical examination (symptomatic arm or hand dysfunction is obligatory).

DETAILED DESCRIPTION:
See Above. Further information in this registration ( Randomized controlled trial (RCT), sample size etc)

ELIGIBILITY:
Inclusion Criteria:

- all patients with a history of a traumatic event to the cervical spine fulfilling the criteria of incomplete cervical spinal cord lesion. -

Exclusion Criteria:

* cognitive impairments
* a preexistent neurologic deficit of arms and/or legs
* psychiatric illness
* significant comorbidity interfering with the indication to perform surgery or not
* use of anticoagulating drugs
* addiction to drugs or alcohol (more than five units daily)
* not speaking Dutch language fluently
* not willing to participate
* participating in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Dutch translation of mJOA | two years post-injury
  functional outcome at two years measured by Dutch translation of mJOA

SECONDARY OUTCOMES:
DASH | two years post-injury
  arm/hand function assessed by the disability of the arm, shoulder and hand questionnaire (DASH)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Bartels, M.D.,Ph.D., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Bartels RH, Hosman AJ, van de Meent H, Hofmeijer J, Vos PE, Slooff WB, Oner FC, Coppes MH, Peul WC, Verbeek AL. Design of COSMIC: a randomized, multi-centre controlled trial comparing conservative or early surgical management of incomplete cervical cord syndrome without spinal instability. BMC Musculoskelet Disord. 2013 Jan 31;14:52. doi: 10.1186/1471-2474-14-52. PMID 23369169